CLINICAL TRIAL: NCT00179478
Title: Controlled High-risk Avonex Multiple Sclerosis Prevention Study in Ongoing Neurologic Surveillance (CHAMPIONS10)
Brief Title: Long Term Study of Avonex Therapy Following a First Attack of Multiple Sclerosis
Acronym: CHAMPIONS10
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Biogen (Industry)
Responsible Party: Principal Investigator, R. Philip Kinkel, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2003P000086; C-850 Extension study (Other: Biogen Inc)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-08

CONDITIONS: Multiple Sclerosis; Optic Neuritis; Transverse Myelitis; Acute Brainstem/Cerebellar Syndrome
Keywords: Multiple sclerosis; Interferon Beta; MRI; Optic neuritis; Transverse Myelitis
MeSH Terms: conditions — Multiple Sclerosis; Optic Neuritis; Myelitis, Transverse; Cerebellar Diseases | interventions — Interferon beta-1a

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Open label study: The outcome committee determined the primary outcome event (the development of Clinically definite MS) without knowledge of original treatment assignment and the central MRI reading center was not aware of original treatment assignments
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Treatment Group (Experimental): Initiation of treatment with Interferon Beta 1a IM once weekly immediately after onset of a first demyelinating syndrome in high risk individuals
  Interventions: Drug: interferon beta 1a 30 ug IM once weekly
- Delayed Treatment Group (Active Comparator): Delayed initiation of of Interferon beta-1a IM once weekly at diagnosis of clinically definite MS, at conclusion of initial CHAMPS study or during long term observation
  Interventions: Drug: interferon beta 1a 30 ug IM once weekly

INTERVENTIONS:
Drug: interferon beta 1a 30 ug IM once weekly — Immediate treatment group refers to those patients who were randomized to the interferon beta 1a 30 ug IM once weekly treatment arm of the original, controlled phase III CHAMPS study; Delayed treatment group refers to those patients who were randomized to the placebo group during the original controlled, phase III CHAMPS study and did not start treatment, if at all, until they completed the CHAMPS study protocol at a later date.

SUMMARY:
The current study is a continuation of the 5 year extension study of the phase III CHAMPS study (see reference). This study was designed to determine if immediate initiation of therapy with Interferon Beta-1a (AVONEX) after a first attack of multiple sclerosis (MS) continues to delay the development of further attacks (CDMS) and the development of neurological disability over a 10 year period of observation. The initial 5 year extension study, called CHAMPIONS5, reported that immediate initiation of interferon Beta-1a (AVONEX) after a first attack of MS continued to delay the development of CDMS and lowered relapse rates compared to delayed initiation of disease modifying treatment (usually with AVONEX) either at the time of a second attack or at the end of the phase III study (24 months). The study was extended to 10 years to determine if these effects are sustained and result in less long term permanent disability.

DETAILED DESCRIPTION:
The CHAMPS study determined that immediate initiation of interferon beta 1a therapy (AVONEX) immediately following a first clinical demyelinating event in high risk patients (i.e. those with at least 2 asymptomatic white matter lesions on cranial MR imaging > 3 mm in diameter or ovoid) delayed the development of clinical definite Multiple Sclerosis (CDMS)(as defined by a second, clinically verifiable attack involving another part of the central nervous system) over 2 years of observation and significantly decreased the development of new or enlarging white matter lesions on MRI over 18 months (see reference). The current study is a long term extension of a cohort of CHAMPS study site and participants. The three main aims of the study are as follows:

1. To determine the long term neurological outcome in patients treated with interferon beta 1a (AVONEX) from onset of a first clinical demyelinating event
2. To determine if immediate initiation of AVONEX therapy (the CHAMPS Avonex treatment group) confers long term benefits compared to delayed initiation of therapy (the CHAMPS placebo group) on the rate of development of CDMS, annualized relapse rates, the development of permanent disability and MR measures of disease activity and progression.
3. To determine predictors of long term disease activity and disability in patients following a first clinical demyelinating event

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in CHAMPS study
* Participation in a study site willing to participate in the CHAMPIONS10 extension study
* Willingness to enroll in the CHAMPIONS 10 extension
* Willingness to sign informed consent

Exclusion Criteria:

* Discovery of an alternative neurological disorder other than MS as a cause of initial neurological symptoms
* A severe systemic disease with likely mortality within 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2001-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Revere P Kinkel, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (26):
- United States (20):
  - MS Treatment Center at Griffin Hospital, Derby, Connecticut
  - Jaeb Center for Health Research, Tampa, Florida
  - MS Center of Atlanta, Atlanta, Georgia
  - Beta Research, Inc, Elk Grove, Illinois
  - University of Iowa College of Medicine, Iowa City, Iowa
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Michigan State University, East Lansing, Michigan
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Jacobs Neurological Institute, Buffalo, New York
  - University of Rochester, Rochester, New York
  - Carolinas Medical Center - MS Center, Charlotte, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - The Neurology Group, Norristown, Pennsylvania
  - Univeristy of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Allegheny Neurological Associates, Pittsburgh, Pennsylvania
  - Univeristy of Texas Houston Health Science Center, Houston, Texas
  - Virginia Commonwealth University/Medical College of Virginia, Richmond, Virginia
  - Neurological Associates, Inc., Richmond, Virginia
  - Marshfield Clinic, Marshfield, Wisconsin
- Canada (6):
  - Vancouver Hospital Health Sciences Centre, Vancouver, British Columbia
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Ottawa General Hospital, Ottawa, Ontario
  - University of Toronto - St. Michael's Hospital, Toronto, Ontario
  - Hospital Notre Dame, Montreal, Quebec
  - Montreal Neurological Institute, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jacobs LD, Beck RW, Simon JH, Kinkel RP, Brownscheidle CM, Murray TJ, Simonian NA, Slasor PJ, Sandrock AW. Intramuscular interferon beta-1a therapy initiated during a first demyelinating event in multiple sclerosis. CHAMPS Study Group. N Engl J Med. 2000 Sep 28;343(13):898-904. doi: 10.1056/NEJM200009283431301. PMID 11006365
- [Background] Kinkel RP, Kollman C, O'Connor P, Murray TJ, Simon J, Arnold D, Bakshi R, Weinstock-Gutman B, Brod S, Cooper J, Duquette P, Eggenberger E, Felton W, Fox R, Freedman M, Galetta S, Goodman A, Guarnaccia J, Hashimoto S, Horowitz S, Javerbaum J, Kasper L, Kaufman M, Kerson L, Mass M, Rammohan K, Reiss M, Rolak L, Rose J, Scott T, Selhorst J, Shin R, Smith C, Stuart W, Thurston S, Wall M; CHAMPIONS Study Group. IM interferon beta-1a delays definite multiple sclerosis 5 years after a first demyelinating event. Neurology. 2006 Mar 14;66(5):678-84. doi: 10.1212/01.wnl.0000200778.65597.ae. Epub 2006 Jan 25. PMID 16436649
- [Background] Kinkel RP, Dontchev M, Kollman C, Skaramagas TT, O'Connor PW, Simon JH; Controlled High-Risk Avonex Multiple Sclerosis Prevention Study in Ongoing Neurological Surveillance Investigators. Association between immediate initiation of intramuscular interferon beta-1a at the time of a clinically isolated syndrome and long-term outcomes: a 10-year follow-up of the Controlled High-Risk Avonex Multiple Sclerosis Prevention Study in Ongoing Neurological Surveillance. Arch Neurol. 2012 Feb;69(2):183-90. doi: 10.1001/archneurol.2011.1426. Epub 2011 Oct 10. PMID 21987393
- [Background] Simon JH, Kinkel RP, Kollman C, O'Connor P, Fisher E, You X, Hyde R; CHAMPIONS Investigators Group. Ten-year follow-up of the 'minimal MRI lesion' subgroup from the original CHAMPS Multiple Sclerosis Prevention Trial. Mult Scler. 2015 Apr;21(4):415-22. doi: 10.1177/1352458514547407. Epub 2014 Oct 24. PMID 25344370
- [Background] Kinkel RP, Laforet G, You X. Disease-related determinants of quality of life 10 years after clinically isolated syndrome. Int J MS Care. 2015 Jan-Feb;17(1):26-34. doi: 10.7224/1537-2073.2013-041. PMID 25741224

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in the CHAMPIONS 5 year extension study were offered participation in the 10 year extension if their study site participated in the 10 year extension. Study arms were already establish at the onset of CHAMPIONS 10 extension
Period: Overall Study
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Started | 81 | 74
Completed | 68 | 59
Not Completed | 13 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Treatment Group | Delayed Treatment Group | Total
Number analyzed (Participants) | 81 | 74 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (7) | 34 (7) | 34 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 53 | 113
  Male | 21 | 21 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 72 | 69 | 141
  Race/Ethnicity: Non White | 9 | 5 | 14
Family History of MS [Count of Participants; unit: Participants] | 12 | 7 | 19
Brainstem/Cerebellar at onset [Count of Participants; unit: Participants] | 21 | 19 | 40
Optic neuritis at onset [Count of Participants; unit: Participants] | 40 | 38 | 78
Spinal cord syndrome at onset [Count of Participants; unit: Participants] | 20 | 17 | 37
EDSS < 2.0 at onset [Count of Participants; unit: Participants] — Expanded Disability Status Scale (EDSS) is an ordinal measure of Neurological disability in Multiple Sclerosis ranging from 0-10 (0.5 increments) where 0 is normal and 10 is death from MS
  Participants | 47 | 55 | 102
EDSS 2.0-2.5 at onset [Count of Participants; unit: Participants] | 24 | 15 | 39
EDSS > 2.5 at onset [Count of Participants; unit: Participants] | 10 | 4 | 14
Median T2 lesion # at onset [Median (Inter-Quartile Range); unit: lesion counts] | 13 [8 to 22] | 13 [9 to 20] | 13 [8 to 21]
Median T2 lesion vol at onset [Median (Inter-Quartile Range); unit: mm^3] | 2063 [1003 to 4945] | 1774 [786 to 4883] | 1930 [918 to 4945]
Gad enhancing lesions at onset [Count of Participants; unit: Participants] | 26 | 17 | 43

OUTCOME MEASURES:

1. Primary Outcome: Rate of Development of Clinical Definite Multiple Sclerosis (CDMS) Over 10 Years
Description: Percent cumulative probability of developing CDMS over 10 years . CDMS was defined as the development of new visual or neurological symptoms discrete from the patients initial event with objective findings on examination.
Time Frame: 10 years
Measure: Number (95% Confidence Interval); unit: Percent cumulative probability
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 81 | 74
Percent cumulative probability | 58 [48 to 68] | 69 [61 to 78]
Statistical Analysis 1: Comparison: Immediate Treatment Group vs Delayed Treatment Group; Test type: Superiority; p = 0.001, Regression, Cox — Based on adjusted Hazard Ratio (HR); HR adjusted for age, onset event type, baseline brain MRI T2 lesion and number and baseline number of gad enhancing lesions

2. Secondary Outcome: Annualized Relapse Rate
Description: annualized # of relapses between years 0 and 10
Time Frame: 10 years
Population: Analysis only in 10 year completers
Measure: Mean (Standard Deviation); unit: annualized relapses per year
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 68 | 59
annualized relapses per year | 0.16 (0.18) | 0.33 (0.41)
Statistical Analysis 1: Comparison: Immediate Treatment Group vs Delayed Treatment Group; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance was a p value less than 0.01

3. Secondary Outcome: Number of Participants With an EDSS > 3.5 at Study Completion
Description: The EDSS is an ordinal scale of neurological impairment in Multiple Sclerosis with a range of 0 to 10 with 0.5 increments. A score of 0 is normal and 10 is death from MS. Scores from 1 to 3.5 are considered mild impairment , 4.0 to 6.5 is moderate and greater than 6.5 is severe impairment.
Time Frame: 10 years
Population: Numbers of patients completing 10 year evaluations
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 68 | 59
Participants | 7 | 5
Statistical Analysis 1: Comparison: Immediate Treatment Group vs Delayed Treatment Group; Test type: Superiority; p = 0.61, Fisher Exact — a priori threshold for statistical significance was a p value < 0.01

4. Secondary Outcome: The Number of New or Enlarging MRI T2 Lesions at 10 Years
Description: These are counts of new or significantly enlarged lesions over 10 years on brain MRI reflecting interval radiographic disease activity
Time Frame: 10 years
Population: Analysis restricted to those participants with MRI scans able to evaluate at 10 years
Measure: Median (Inter-Quartile Range); unit: # of new or enlarging T2 lesions
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 55 | 55
# of new or enlarging T2 lesions | 5 [1 to 12] | 7 [3 to 17]
Statistical Analysis 1: Comparison: Immediate Treatment Group vs Delayed Treatment Group; Test type: Superiority; p = 0.50, Fisher Exact — a priori threshold for statistical significant was a p value less than 0.01

ADVERSE EVENTS:
Time Frame: Non serious and serious adverse events were not recorded during this extension study. For this study (n=155) only information on mortality was collected and categorized.
Groups:
- All Study Participants: All patients in the study were receiving the same FDA approved treatment, interferon beta 1a IM once weekly (AVONEX), which they received commercially through their insurance coverage. No AEs were collected and any serious AEs that occurred, would have been reported to the manufacturer (Biogen). We collected information on all cause mortality on the cohort of 155 patients who continued in the 10 year extension study. This was done as an additional outcome measure since we anticipated that there may be deaths due to the primary disease (MS) over a period of observation as long as 10 years.
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 2/155
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
selective attrition of patients with greater levels of disease activity may have occurred in this long term extension study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No